CLINICAL TRIAL: NCT06095583
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Regional Phase III Clinical Study of Toripalimab Alone or in Combination With Tifcemalimab (JS004/TAB004) as Consolidation Therapy in Patients With Limited-Stage Small Cell Lung Cancer Without Disease Progression Following Chemoradiotherapy
Brief Title: Phase 3 Study of Toripalimab Alone or in Combination With Tifcemalimab as Consolidation Therapy in Patients With Limited-stage Small Cell Lung Cancer (LS-SCLC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS004-008-III-SCLC
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Limited-stage Small Cell Lung Cancer (LS-SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — toripalimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental group A (Experimental): Tifcemalimab (200 mg intravenous infusion [IV]) and toripalimab (240 mg IV)
  Interventions: Drug: Tifcemalimab injection; Drug: toripalimab injection
- Experimental group B (Experimental): Placebo for tifcemalimab (IV) and toripalimab (240 mg IV)
  Interventions: Drug: toripalimab injection; Drug: Placebo for Tifcemalimab
- Placebo group C (Placebo Comparator): Placebos for both tifcemalimab and toripalimab (IV)
  Interventions: Drug: Placebo for Tifcemalimab; Drug: Placebo for toripalimab

INTERVENTIONS:
Drug: Tifcemalimab injection — 200mg once every 3weeks
  Arms: Experimental group A
Drug: toripalimab injection — 240mg once every 3 weeks
  Arms: Experimental group A; Experimental group B
Drug: Placebo for Tifcemalimab — every 3weeks
  Arms: Experimental group B; Placebo group C
Drug: Placebo for toripalimab — every 3weeks
  Arms: Placebo group C

SUMMARY:
The Study is a Phase 3, randomized, three-arm, double-blind, placebo-controlled, multi-regional clinical research study to evaluate the safety and efficacy use of toripalimab alone or in combination with tifcemalimab as consolidation therapy in patients with limited-stage small cell lung cancer without disease progression following chemoradiotherapy.

Tifcemalimab is a monoclonal antibody against B and T lymphocyte attenuator (BTLA). Toripalimab is a monoclonal antibody against programmed death protein-1 (PD-1). Neither drug is approved for treatment of This combination regimen is investigational in limited stage-small cell lung cancer in any country.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be enrolled:

1. Male or female with age ≥ 18 years old at the time of informed consent.
2. Histologically or cytologically confirmed LS-SCLC using the Veteran's Administration Lung Study Arm (VALSG) staging criteria (Appendix 3). Patients with TNM Stage I or II disease per AJCC 8th edition must be medically inoperable (as determined by the Investigator) or the patient must refuse surgery.
3. Received CRT defined as: (1) 4 cycles of chemotherapy consisting of carboplatin or cisplatin and intravenously administered etoposide; (2) a total radiation dose of 60-66 Gy for the standard once daily (QD) radiotherapy regimen or 45 Gy for the hyperfractionated twice daily (BID) radiotherapy regimen; (3) Patients must begin investigational interventions within 42 days of the last dose of chemotherapy.
4. Patients must have achieved a complete response (CR), partial response (PR), or stable disease (SD) after receiving curative platinum-based CRT and must not have developed progressive disease (PD) prior to study entry.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-1 .
6. Adequate organ function
7. Female patients of childbearing potential and male patients whose partners are women of childbearing age.
8. Voluntarily agree to participate in the study, sign the informed consent form, and agree to comply with all study and follow-up procedures.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria.

1. Mixed SCLC and non-small cell lung cancer (NSCLC).
2. Received sequential chemoradiotherapy for LS-SCLC.
3. Failure to recover from toxicity of prior anticancer therapy to Common Terminology Criteria for Adverse Events (CTCAE) Grade ≤ 1 (except alopecia) or levels specified in the inclusion/exclusion criteria, whichever is more severe.
4. Patients with active autoimmune disease, history of autoimmune disease.
5. History of immunodeficiency, including HIV seropositivity, other acquired congenital immunodeficiency diseases, or a history of organ transplantation or allogeneic bone marrow transplantation.
6. History of confirmed or suspected interstitial lung disease or pneumonitis (except for Grade 1 radiation pneumonitis not treated with corticosteroids).
7. The presence of active hepatitis B (HBV DNA ≥ 500 IU/mL), hepatitis C (hepatitis C antibodies positive and HCV-RNA higher than the lower limit of detection of the analytical method).
8. Any other malignancy diagnosed prior to the first dose of investigational intervention, except those with a low risk for the development of metastases (5-year survival rate > 90%), such as adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or breast, or adequately treated localized prostate cancer.
9. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 3years
  To compare and evaluate the efficacy of tifcemalimab and toripalimab (Arm A) versus placebo (Arm C) as consolidation therapy after chemoradiotherapy (CRT) for patients with LS-SCLC as measured by OS
OS | up to 3years
  To compare and evaluate the efficacy of toripalimab (Arm B) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLC as measured by OS"
Progression-free survival (PFS) | up to 2years
  To compare and evaluate the efficacy of tifcemalimab and toripalimab (Arm A) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLC as measured by Blinded Independent Review Committee (BIRC)-assessed PFS.
Progression-free survival (PFS) | up to 2years
  To compare and evaluate the efficacy of toripalimab (Arm B) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLC as measured by OS and BIRC-assessed PFS.

SECONDARY OUTCOMES:
PFS | up to 2years
  To compare and evaluate the efficacy of tifcemalimab and toripalimab (Arm A) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLC as measured by Investigator-assessed PFS
1-year OS rate | up to 1year
  To compare and evaluate the efficacy of tifcemalimab and toripalimab (Arm A) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLC as measured by 1-year OS rate
2-year OS rate | up to 2 years
  To compare and evaluate the efficacy of tifcemalimab and toripalimab (Arm A) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLC as measured by 2-year OS rate
objective response rate (ORR) | up to 2 years
  To compare and evaluate the efficacy of tifcemalimab and toripalimab (Arm A) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLC as measured by ORR
disease control rate (DCR) | up to 2 years
  To compare and evaluate the efficacy of tifcemalimab and toripalimab (Arm A) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLC as measured by DCR
duration of response (DoR) | up to 2years
  To compare and evaluate the efficacy of tifcemalimab and toripalimab (Arm A) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLC as measured by DoR
PFS | up to 2 years
  To compare and evaluate the efficacy of toripalimab (Arm B) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLS as measured by Investigator-assessed PFS
1 year OS rate | up to 1 years
  To compare and evaluate the efficacy of toripalimab (Arm B) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLS as measured by 1-year OS rate
2 year OS rate | up to 2 years
  To compare and evaluate the efficacy of toripalimab (Arm B) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLS as measured by 2-year OS rate
ORR | up to 2 years
  To compare and evaluate the efficacy of toripalimab (Arm B) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLS as measured by ORR
DCR | up to 2 years
  To compare and evaluate the efficacy of toripalimab (Arm B) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLS as measured by DCR
DoR | up to 2 years
  To compare and evaluate the efficacy of toripalimab (Arm B) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLS as measured by DoR
safety | up to 2 years
  To compare and evaluate the safety of tifcemalimab and toripalimab (Arm A) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLC as measured by the incidence of adverse events (Percentage of participants with treatment-related adverse events as assessed by CTCAEv5.0.) and abnormal laboratory parameters.
safety | up to 2 years
  To compare and evaluate the safety of toripalimab (Arm B) versus placebo (Arm C) as consolidation therapy after CRT for patients with LS-SCLC as measured by the incidence of adverse events (Percentage of participants with treatment-related adverse events as assessed by CTCAEv5.0.) and abnormal laboratory parameters.

CONTACTS AND LOCATIONS:
Locations (156):
- United States (29):
  - Banner MD Anderson Cancer Center, Goodyear, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - Genesis Cancer and Blood Institute (Hot Springs, AR), Hot Springs, Arkansas
  - SCRI Nashville, Davis, California
  - Zangmeister Cancer Center (Columbus, OH), Los Angeles, California
  - Los Angeles Hematology Oncology, Los Angeles, California
  - University of Southern California Norris Comprehensive Cancer, Los Angeles, California
  - Florida Cancer Specialists Pan Handle, Fort Myers, Florida
  - Florida Cancer Specialists South, Fort Myers, Florida
  - USA029 University of Miami Sylvester Comprehensive Cancer Center 1550 NW 10th Avenue 33173 Miami FL Ikpeazu Chukwuemeka N, Miami, Florida
  - Mid-Florida Hematology Oncology, Orange City, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Marietta, Georgia
  - Norton Cancer Institute, Downtown, Multidisciplinary Clinic, Louisville, Kentucky
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Dana Farber Cancer Institute-Hematology/Oncology, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - North Shore Hematology Oncology Associates DBA NY Cancer and Blood Specialists, New York, New York
  - University of Stony Brook, Stony Brook, New York
  - Toledo Clinic Cancer Center - Toledo, Toledo, Ohio
  - Oncology Associates Of Oregon, P.C., Eugene, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Millennium Physicians - Oncology, Houston, Texas
  - Texas Oncology, P.A. - Oncology, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Belgium (5):
  - Algemeen Ziekenhuis Klina, Antwerp
  - Grand Hôpital de Charleroi - Site Notre-Dame, Charleroi
  - AZ Groeningen, Kortrijk
  - Jessa Ziekenhuis - Campus Virga Jesse, Limbourg
  - CHU UCL Namur - Site Sainte-Elisabeth, Namur
- China (31):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital & Institute, Jinan, Shandong
  - Anyang Tumor Hospital, Anyang
  - Beijing Cancer Hospital, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - Sichuan cancer hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Peking University Shenzhen Hospital, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou
  - No. 1 Bandong Road, Gongshu District, Hangzhou, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Ustc, Hefei
  - Henan Cancer Hospital, Henan
  - Affiliated Hospital of Jining Medical University, Jining
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Liaoning cancer hospital, Shenyang
  - Shanxi Cancer hospital, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Hubei Cancer Hospital (Hubei Cancer Research Institute), Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - General Hospital of Ningxia Medical University, Yinchuan
- France (12):
  - Centre Hospitalier Universitaire D Angers, Angers
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Intercommunal De Créteil, Créteil
  - CHU de Grenoble, Grenoble
  - Centre Leon Berard - departement d'oncologie medicale, Lyon
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Hopital Arnaud De Villeneuve - Oncologie/Pneumologie, Montpellier
  - Hopital Haut-Leveque - Maladies respiratoires, Pessac
  - Chu Hôpitaux De Rouen, Rouen
  - Institut de Cancérologie de l'Ouest (ICO), Saint-Herblain
  - Chru De Tours, Tours
  - Institut Gustave Roussy, Villejuif
- Georgia (8):
  - "TIM - Tbilisi Institute of Medicine" LTD, Tbilisi
  - ICO-Institute of Clinical Oncology - Hospital, Tbilisi
  - ISR-GEO Med Res Clin Healthycore, Tbilisi
  - LTD "Israel-Georgian Medical Research Clinic Healthycore", Tbilisi
  - LTD "New Hospitals", Tbilisi
  - Ltd New Hospitals, Tbilisi
  - Multprofil Clinic Consilium Medulla, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi
- Germany (6):
  - Evangelische Lungenklinik Berlin, Berlin
  - Klinikum Esslingen GmbH Klinik für Kardiologie, Angiolgie und Pneumolgoie, Esslingen am Neckar
  - Univeristätsklinikum Giessen und Marburg GmbH, Giessen
  - Klinikum Kassel GmbH Klinik für Onkologie uind Hämatologie- Onkologisches Studiensekretariat, Kassel
  - Gemeinschaftspraxis fuer Haematologie und Onkologie, Münster
  - Universitätsklinikum Regensburg, Regensburg
- Italy (9):
  - PO G. Rodolico, AOU Policlinico-Vittorio Emanuele Catania, Catania
  - Istituto Romagnolo per lo Studio dei Tumori (IRST) Dino Amadori IRCCS, Cesena
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliero-Universitaria di Modena, Policlinico di Mod, Modena
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli, Napoli
  - Iov, Irccs, Padua
  - IRCCS Policlinico San Matteo, Università degli studi di Pavia, Pavia
  - AO S. Camillo-Forlanini, Roma
  - Regina Elena, Istituto Nazionale dei Tumori, IFO, IRCCS Feasibility survey: PO di Livorno, AUSL Toscana Nord Ovest, SST, Roma
- Netherlands (4):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Rijnstate Ziekenhuis, Arnhem
  - Erasmus Medisch Centrum, Rotterdam
  - Isala Klinieken Zwolle, Zwolle
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - SPZOZ MSWiA z Warminsko-Mazurskim Centrum Onkologii, Olsztyn
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii im. E. i J. Zeylandow, Poznan
  - Instytut Gruzlicy i Chorob Pluc, Warsaw
- Romania (6):
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj-Napoca, Cluj-Napoca
  - Medisprof, Cluj-Napoca
  - Centrul de Oncologie Sf. Nectarie, Craiova
  - Oncolab, Craiova
  - Radiotherapy Center Cluj, Floreşti
  - Oncomed, Timișoara
- South Korea (3):
  - Chungbuk National University Hospital, Cheonju
  - Seoul National University Bundang Hospital, Seongnam
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (15):
  - Centro Oncológico de Galicia, A Coruña
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Dexeus Grupo Quironsalud, Barcelona
  - C.H. Provincial de Castellón, Castellon
  - Complejo Hospitalario de Jaén, Jaén
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario Universitario de Orense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario Virgen De La Macarena, Seville
  - Hospital Arnau De Vilanova De Valencia, Valencia
  - Hospital Universitario Y Politécnico La Fe, Valencia
  - H.C.U.Lozano Blesa, Zaragoza
- Taiwan (11):
  - Taipei Veterans General Hospital, Taipei City, Taipei
  - No.123,DAPI Rd. Niaosong Dist, Kaohsiung City 83301 Taiwan, R.O.C., Kaohsiung City
  - China Medical University Hospital - Internal Medicine - Taichung, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Hospital, Liouying - Department of Oncology, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital - Internal Medicine, Taipei
  - Taipei Medical University - Shuang Ho Hospital, Taipei
  - Taipei Medical University - Taipei Medical University Hospital, Taipei
  - Taipei Medical University - WanFang Hospital - Hematology and Oncology, Taipei
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (13):
  - Ankara City Hospital, Ankara
  - Ankara Liv Hospital, Ankara
  - Gulhane Training and Research Hospital - Medical Oncology, Ankara
  - Memorial Ankara Hospital, Ankara
  - Trakya University Medical Faculty, Edirne
  - Bakirköy Dr. Sadi Konuk Eğitim ve Araştirma Hastanesi - Oncology, Istanbul
  - Istanbul Goztepe Prof. Dr. Suleyman Yalcin City Hospital - Medical Oncology, Istanbul
  - Ege University Medical Faculty - Pulmonary, Izmir
  - İzmir Ekonomi Üniversitesi Medical Point İzmir Hastanesi, Izmir
  - Katip Celebi University Ataturk Research and Training Hospit, Izmir
  - Kocaeli University Research and Practice Hospital, Kocaeli
  - Necmettin Erbakan University Meram, Konya
  - Inonu University Turgut Ozal Medical Center, Malatya

IPD SHARING:
Plan to Share IPD: No